CLINICAL TRIAL: NCT05696509
Title: Influence of Anesthetics on Clinical Outcome in Mitral and Aortic Valve Replacement in Adults: a Randomized Clinical Trial
Brief Title: Influence of Anesthetics on Clinical Outcome in Mitral and Aortic Valve Replacement in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Bekzat Baiterek, 2nd year doctoral student, anesthesiologist, resuscitator, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AMU3
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Mitral Valve Insufficiency; Aortic Valve Insufficiency
Keywords: clinical outcome; sevoflurane; isoflurane; propofol; Mitral Valve Insufficiency; Aortic Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency; Aortic Valve Insufficiency | interventions — Propofol; Anesthesia; Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Other): Anesthetic
  Interventions: Drug: Propofol
- Isofluran (Other): Anesthetic
  Interventions: Drug: Isoflurane
- Sevofluran (Other): Anesthetic
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 4-6 mg/kg/h intravenously on a perfusor.
  Other Names: Anesthesia
  Arms: Propofol
Drug: Isoflurane — Isoflurane was used as an anaesthetic in a dose of - 1.1-1.2 MAC
  Other Names: Anesthesia
  Arms: Isofluran
Drug: Sevoflurane — sevoflurane was used as an anaesthetic in a dose of - 1.7-1.9 MAC
  Other Names: Anesthesia
  Arms: Sevofluran

SUMMARY:
Abstract Anaesthetic support for cardiac surgery significantly influences the course of the intraoperative period and the success of the postoperative period. Total intravenous anaesthesia and inhalation anaesthesia are the traditional methods of anaesthesia in cardiac surgery. However, there are few studies assessing the effectiveness of surgical aggression protection in cardiac surgery.

Objectives: To study the effect of anesthetics on clinical outcome after mitral and aortic valve replacement in adults.

Methods. The data of 75 patients operated in the Cardiosurgery Department of the Medical Center Hospital of the Presidential Administration of the Republic of Kazakhstan were included in the study. All patients underwent mitral, aortic valve replacement/plasty under cardiopulmonary bypass (CPB) conditions.

All patients were divided into 3 groups according to the type of anaesthesia: the first (1) group patients anaesthetised with propofol (P), the second group with sevoflurane (S), and the last one is with isoflurane (I).

To maintain anaesthesia in Group 1 propofol was used as anaesthetic in a dose of 6 mg/kg/h intravenously on perfusion. In Group 2 the anaesthetic used was sevoflurane in a dose of 1.7-1.9 MAC. Group 3 used isoflurane in the dose of 1.1-1.2 MAC as anaesthetic. Statistical analysis was done by the method of single factor analysis of variance and Kruskal Wallis criterion.

DETAILED DESCRIPTION:
This study includes data from 90 patients operated in the Cardiosurgery Department of the Medical Center Hospital of the Presidential Administration of the Republic of Kazakhstan were included in the study. All patients underwent mitral, aortic valve replacement/plasty under cardiopulmonary bypass (CPB) conditions. This research work was conducted between 2020 and 2022. To calculate the sample size, the investigators used the formula n=t2*D*N/confidence interval*N+t2*α, which will allow to identify the static significance of the study.

All patients were divided into 3 groups according to the type of anaesthesia: the first (1) group patients anaesthetised with propofol (P), the second group with sevoflurane (S), and the last one is with isoflurane (I).

The study was conducted in 5 stages:

1. Initial haemodynamic parameters and oxygen transport function of the patient's blood before anaesthesia were determined;
2. After tracheal intubation;
3. Before the CPB;
4. After the CPB;
5. The post-operative period until the patient is transferred to the specialized department.

Before induction into anaesthesia, haemodynamic monitoring was started on admission to the operating theatre using a Nihon Kohden monitor (Japan). The right radial artery was catheterised for invasive monitoring of systemic arterial pressure and arterial blood sampling, and a catheter was then inserted into the central jugular vein (under ultrasound machine control) and guided into the right atrium for mixed venous blood sampling.

Cardiac stroke volume was determined by transthoracic echocardiography (CS=end diastolic volume - end systolic volume). Cardiac output (CO=CS x heart rate), cardiac index (CI=CO/body surface area) were determined. the investigators determined blood oxygen content using the formula CaO2 (arterial ABB) and CvO2 (central mixed venous ABB) = [(1.34 × Hb × SO2) + (PO2 × 0.031)] / 100. Arteriovenous difference = CaO2-CvO2. Oxygen delivery was determined using the formula (DO2 = CI* CaO2). Oxygen consumption (VO2 = Cardiac index (CI)*AVD or VO2 = CO × (CaO2 - CvO2) ~ CO × Hb × 1.34 × (SaO2 - SvO2) / 100).

In the second stage, after tracheal intubation, indirect calorimetry was used to determine VO2, energy expenditure during anaesthesia using a Spirometry device (Oxford, UK), which was connected to an endotracheal tube and continuously showed oxygen demand and energy expenditure. A transesophageal echocardiography sensor was used to determine cardiac output. Additionally, the cardiac output was determined by Fick's formula. The same tests (cardiac output, cardiac index, consumption, oxygen delivery, energy expenditure) were performed in the third and fourth stages of anaesthesia. In the last stage, the consumption of muscle relaxants and opioid analgesics was calculated to assess the pharmaco-efficiency of anaesthetics. The time of extubation and the time of transfer of the patient to the specialized department were determined.

All patients continued antihypertensive medication both before and on the day of surgery to prevent the development of withdrawal syndrome and to reduce the risk of perioperative myocardial ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* The age is between 40-60 years old;
* Mitral valve insufficiency grade 3-4;
* Aortic valve insufficiency grade 3-4;
* Participants of both sexes will be included in the study;
* Signed informed consent.

Exclusion Criteria:

* pregnancy (risk to the baby and the mother)

  * allergenic patients (anaphylactic shock).
  * vulnerable groups.
  * current congestive heart failure;
  * current unstable angina pectoris;
  * preoperative hemodynamic instability, defined as the use of vasopressors;

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
cardiac index | 1 year
  The cardiac stroke (CS) volume was determined by transthoracic echocardiography (CS=end diastolic volume-end systolic volume). There were also determined the cardiac output (CO=CS x heart rate), cardiac index (CI=CO/body surface area).
Oxygen consumption | 1 year
  Oxygen consumption (VO2 = Cardiac index *AVD or VO2 = CO × (CaO2 - CvO2) ~ CB × Hb × 1,34 × (SaO2 - SvO2) / 100), oxygen utilization factor (KYO2) = VO2 / DO2 × 100 = [(CaO2 - CvO2) / CaO2] × 100.
Oxygen delivery | 1 year
  The oxygen delivery was found by formula (DO2 = CI* CaO2)

CONTACTS AND LOCATIONS:
Overall Officials: Alibek Kh Mustafin, Professor, Study Chair — Astana Medical University
Locations (1):
- Bekzat, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
To study the effect of anesthetics on clinical outcome after mitral and aortic valve replacement in adults.